CLINICAL TRIAL: NCT03825939
Title: Evaluating the Use of Tranexamic Acid (TXA) in Total Joint Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patient enrollment due to only one surgeon that was enrolling.
Sponsor: NYU Langone Health (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WUH 592498-2
Record Dates: First submitted 2015-12-23; First posted 2019-02-01 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Blood Loss
Keywords: Total hip arthroplasty; Total knee arthroplasty
MeSH Terms: conditions — Hemorrhage | interventions — Sodium Chloride; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intravenous Tranexamic Acid (Experimental): * 1g TXA administered intravenous piggyback at start of surgery OR
  * 1g TXA administered intravenous piggyback at start and at time of closure of surgery
  Interventions: Drug: Intravenous Tranexamic Acid
- Intravenous Placebo (Placebo Comparator): - IV 0.9% sterile saline
  Interventions: Drug: Intravenous Placebo
- Intravenous Tranexamic Acid followed by Intravenous Placebo (Active Comparator): * 1g TXA administered intravenous piggyback at start of surgery OR
  * 1g TXA administered intravenous piggyback at start and at time of closure of surgery
  * IV 0.9% sterile saline
  Interventions: Drug: Intravenous Placebo; Drug: Intravenous Tranexamic Acid

INTERVENTIONS:
Drug: Intravenous Placebo — IV 0.9% sterile saline
  Other Names: Saline
  Arms: Intravenous Placebo; Intravenous Tranexamic Acid followed by Intravenous Placebo
Drug: Intravenous Tranexamic Acid — 1g TXA IVPB (intravenous piggyback)
  Other Names: Tranexamic Acid
  Arms: Intravenous Tranexamic Acid; Intravenous Tranexamic Acid followed by Intravenous Placebo

SUMMARY:
This research study aims to study the use of tranexamic acid (TXA) in total joint replacement (arthroplasty) of the hip (THR) and knee (TKR).

DETAILED DESCRIPTION:
Tranexamic Acid (TXA) is given to stop or reduce heavy bleeding. It works by stopping clots from breaking down and by decreasing unwanted bleeding. It is used in many types of surgeries to help reduce surgical complications such as blood loss and blood transfusions.

In orthopaedic surgeries, such as in total hip and knee replacements, TXA has been shown to effectively reduce blood loss and transfusion requirements without an increased risk of side effects such as deep venous thrombosis (DVT) or pulmonary embolism (PE). The ability to decrease blood loss is crucial, as other studies have shown that reducing blood loss decreases morbidity and mortality in patients.

Although, many TXA dosing regimens have been studied - all of which have been useful at reducing blood loss and decreasing transfusion requirements - the best TXA dosing regimen and the most cost-effective method of TXA administration for patients have yet to be determined. Moreover, a thorough and rigorous study on the use and effects of topical and intravenous TXA and the effect of TXA on patient outcomes has yet to be conducted.

Therefore, this research study aims to address those concerns in order to understand how best to use TXA to reduce surgical complications in patients undergoing total joint replacements.

ELIGIBILITY:
Inclusion Criteria

* All patients 18 years and older who are already scheduled for primary total joint arthroplasty of the hip or knee

Exclusion Criteria for IV TXA administration

* Cardiac stent or ischemic stroke or coronary artery bypass graft (CABG)
* If patient is on anticoagulant, patient must have documented approval from a cardiologist that patient can be removed from anticoagulant for total joint arthroplasty procedure
* Renal impairment defined as serum Cr > 1.5 or Cr Clearance < 50 mL/min
* Severe ischemic heart disease
* Color blindness or problems with color vision

Criteria for Use of Topical TXA

* Topical TXA can be used in any patient meeting one of the exclusion criteria for IV TXA administration (Section 5.3b) as there is minimal systemic absorption with topical TXA

Absolute Exclusion Criteria

* History of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Known congenital thrombophilia
* History of thromboembolic or vascular disease
* Disseminated intravascular coagulation (DIC)
* History of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Koenig, M.D., Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Pedersen AB, Mehnert F, Overgaard S, Johnsen SP. Allogeneic blood transfusion and prognosis following total hip replacement: a population-based follow up study. BMC Musculoskelet Disord. 2009 Dec 29;10:167. doi: 10.1186/1471-2474-10-167. PMID 20040083
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Panteli M, Papakostidis C, Dahabreh Z, Giannoudis PV. Topical tranexamic acid in total knee replacement: a systematic review and meta-analysis. Knee. 2013 Oct;20(5):300-9. doi: 10.1016/j.knee.2013.05.014. Epub 2013 Jun 28. PMID 23815893
- [Background] Orpen NM, Little C, Walker G, Crawfurd EJ. Tranexamic acid reduces early post-operative blood loss after total knee arthroplasty: a prospective randomised controlled trial of 29 patients. Knee. 2006 Mar;13(2):106-10. doi: 10.1016/j.knee.2005.11.001. Epub 2006 Feb 17. PMID 16487712
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Niskanen RO, Korkala OL. Tranexamic acid reduces blood loss in cemented hip arthroplasty: a randomized, double-blind study of 39 patients with osteoarthritis. Acta Orthop. 2005 Dec;76(6):829-32. doi: 10.1080/17453670510045444. PMID 16470437
- [Background] Tanaka N, Sakahashi H, Sato E, Hirose K, Ishima T, Ishii S. Timing of the administration of tranexamic acid for maximum reduction in blood loss in arthroplasty of the knee. J Bone Joint Surg Br. 2001 Jul;83(5):702-5. doi: 10.1302/0301-620x.83b5.11745. PMID 11476309
- [Background] Alvarez JC, Santiveri FX, Ramos I, Vela E, Puig L, Escolano F. Tranexamic acid reduces blood transfusion in total knee arthroplasty even when a blood conservation program is applied. Transfusion. 2008 Mar;48(3):519-25. doi: 10.1111/j.1537-2995.2007.01564.x. Epub 2007 Dec 7. PMID 18067499
- [Background] Camarasa MA, Olle G, Serra-Prat M, Martin A, Sanchez M, Ricos P, Perez A, Opisso L. Efficacy of aminocaproic, tranexamic acids in the control of bleeding during total knee replacement: a randomized clinical trial. Br J Anaesth. 2006 May;96(5):576-82. doi: 10.1093/bja/ael057. Epub 2006 Mar 10. PMID 16531440
- [Background] Chang CH, Chang Y, Chen DW, Ueng SW, Lee MS. Topical tranexamic acid reduces blood loss and transfusion rates associated with primary total hip arthroplasty. Clin Orthop Relat Res. 2014 May;472(5):1552-7. doi: 10.1007/s11999-013-3446-0. Epub 2014 Jan 3. PMID 24385043
- [Background] Martin JG, Cassatt KB, Kincaid-Cinnamon KA, Westendorf DS, Garton AS, Lemke JH. Topical administration of tranexamic acid in primary total hip and total knee arthroplasty. J Arthroplasty. 2014 May;29(5):889-94. doi: 10.1016/j.arth.2013.10.005. Epub 2013 Oct 16. PMID 24238825
- [Background] Georgiadis AG, Muh SJ, Silverton CD, Weir RM, Laker MW. A prospective double-blind placebo controlled trial of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):78-82. doi: 10.1016/j.arth.2013.03.038. Epub 2013 Jul 29. PMID 23906869
- [Background] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on transfusion rate in primary total hip arthroplasty. J Arthroplasty. 2014 Feb;29(2):387-9. doi: 10.1016/j.arth.2013.05.026. Epub 2013 Jun 21. PMID 23790499
- [Background] Gilbody J, Dhotar HS, Perruccio AV, Davey JR. Topical tranexamic acid reduces transfusion rates in total hip and knee arthroplasty. J Arthroplasty. 2014 Apr;29(4):681-4. doi: 10.1016/j.arth.2013.09.005. Epub 2013 Oct 4. PMID 24095586
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Gillette BP, DeSimone LJ, Trousdale RT, Pagnano MW, Sierra RJ. Low risk of thromboembolic complications with tranexamic acid after primary total hip and knee arthroplasty. Clin Orthop Relat Res. 2013 Jan;471(1):150-4. doi: 10.1007/s11999-012-2488-z. PMID 22814857
- [Background] Fu DJ, Chen C, Guo L, Yang L. Use of intravenous tranexamic acid in total knee arthroplasty: a meta-analysis of randomized controlled trials. Chin J Traumatol. 2013;16(2):67-76. PMID 23540893
- [Background] Yang ZG, Chen WP, Wu LD. Effectiveness and safety of tranexamic acid in reducing blood loss in total knee arthroplasty: a meta-analysis. J Bone Joint Surg Am. 2012 Jul 3;94(13):1153-9. doi: 10.2106/JBJS.K.00873. PMID 22623147

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Tranexamic Acid: * 1g TXA administered intravenous piggyback at start of surgery OR
  * 1g TXA administered intravenous piggyback at start and at time of closure of surgery
  Intravenous Tranexamic Acid: 1g TXA IVPB
- Intravenous Tranexamic Acid Followed by Intravenous Placebo: * 1g TXA administered intravenous piggyback at start of surgery OR
  * 1g TXA administered intravenous piggyback at start and at time of closure of surgery
  * IV 0.9% sterile saline
  Intravenous Placebo: IV 0.9% sterile saline
  Intravenous Tranexamic Acid: 1g TXA IVPB
Period: Overall Study
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
Started | 18 | 20 | 14
Completed | 18 | 20 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo | Total
Number analyzed (Participants) | 18 | 20 | 14 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6) | 67.2 (11.4) | 65.2 (12.3) | 65.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 8 | 29
  Male | 8 | 9 | 6 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 18 | 12 | 46
  Other | 2 | 2 | 2 | 6
Pre-operative hemoglobin [Median (Standard Deviation); unit: grams/decileter (g/dl)] | 14.4 (1.5) | 13.6 (1.4) | 13.8 (1.5) | 13.9 (1.5)
Pre-operative hematocrit [Mean (Standard Deviation); unit: percentage of red blood cells] | 43.6 (4.6) | 41.2 (4.2) | 41.2 (4.3) | 42.0 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Required a Blood Transfusion During Surgery
Description: Multiple efforts were made to locate the study data, but were unsuccessful (study was terminated, data was not saved). No study data are available.
Time Frame: operative period (average of 1 hour)
Population: Multiple efforts were made to locate the study data, but were unsuccessful (study was terminated, data was not saved). No study data are available.
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Levels of Hematocrit: Pre-operative to Post-operative
Description: as for outcome 1
Time Frame: Day 3 or 4 post surgery
Population: as for outcome 1
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Length of Hospital Stay
Description: Measured in Days
Time Frame: At Hospital Discharge
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
Number analyzed (Participants) | 18 | 20 | 14
Days | 3 [3 to 3] | 3 [2.5 to 3] | 3 [2 to 4]

4. Secondary Outcome: Estimated Blood Loss During Surgery
Description: Surgeon estimated blood loss
Time Frame: Operative period (an average of 1 hour)
Population: as for outcome 1
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Hemoglobin: Pre-operative to Post-operative
Description: Measured in grams/deciliter
Time Frame: Day 3 or 4 post surgery
Population: as for outcome 1
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Walking Distance Post Total Joint Arthroplasty of the Hip
Description: Walking distance (feet) will be assessed and documented throughout the hospital stay
Time Frame: 4 Days
Population: as for outcome 1
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Multiple efforts were made to locate the study data, but were unsuccessful (study was terminated, data was not saved). No study data are available.
Arm/Group | Intravenous Tranexamic Acid | Intravenous Placebo | Intravenous Tranexamic Acid Followed by Intravenous Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes